CLINICAL TRIAL: NCT07166562
Title: Pulse Pressure Variation During Forced Inspiratory Breathing Could Predict Post-Induction Hypotension in Elderly Patients: A Prospective, Observational Study
Brief Title: PPV for Predicting PIH in the Elderly
Acronym: PPVfi-PIH
Status: Not yet recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: LYF20240327
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hypotension on Induction
Keywords: Post-induction Hypotension; Pulse Pressure Variation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this observational study is to investigate the predictive power of pulse pressure variability during forced inhalation（PPVfi） on the occurrence of hypotension in elderly patients after induction of general anesthesia. The main question it aims to answer is:

Can the PPVfi predict the occurrence of hypotension in elderly patients after induction of general anesthesia? By recording the PPV of patients during forced inhalation before anesthesia induction, with the incidence of hypotension as the state variable and PPV as the test variable, the area under the ROC curve was calculated to determine the optimal threshold, sensitivity, and specificity of PPV.

DETAILED DESCRIPTION:
Post-induction hypotension(PIH) usually refers to the hypotension that occurs during the period from anesthesia induction to skin incision, which often occurs during general anesthesia induction. During this period, anesthesiologists may delay the identification and management of hypotension induced by general anesthesia due to their focus on airway management or invasive procedures. Although hypotension usually lasts for a short period of time and can be corrected through fluid replacement and/or medication, there are still studies suggesting that PIH may be associated with adverse postoperative outcomes such as myocardial injury, stroke, and acute kidney injury. Research on predicting PIH both domestically and internationally has focused on evaluating preoperative volume status and autonomic nervous system function. The main indicators for assessing volume responsiveness include pulse pressure variability（PPV）, stroke variability, pulse variability index, perfusion index, etc. Studies have shown that the sensitivity and specificity of pulse pressure variability in identifying PIH are 86% and 86.2%, respectively. In recent years, scholars have proposed that PPV during forced inspiratory breathing (PPVfi) can be used to evaluate patients' volume responsiveness. However, existing research on predicting PIH with pulse pressure variability is mostly focused on middle-aged and young people. However, being over 50 years old is one of the high-risk factors for hypotension after anesthesia induction, and the elderly population has a greater risk of developing hypotension. This study is a non interventional observational prospective study that explores the prediction of hypotension in elderly patients after induction of general anesthesia by exploring the PPV. It helps anesthesiologists to identify and intervene in hypotension after induction of general anesthesia in advance, reducing the occurrence of adverse outcomes after general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification ≤ Grade III;Age ≥ 65 years old; Elective surgery; Patients who require invasive arterial blood pressure monitoring during surgery.

Exclusion Criteria:

* Presence of moderate or severe systemic diseases, such as heart failure, arrhythmias, valvular heart disease, pulmonary hypertension, severe pulmonary diseases (e.g., chronic obstructive pulmonary disease (COPD), asthma, bronchiectasis), endocrine disorders, etc.;Preoperative systolic blood pressure (SBP) ≥160 mmHg, mean arterial pressure (MAP) ≥110 mmHg, or heart rate (HR) ≥120 beats per minute;Patients with comorbid psychiatric or neurological disorders, or communication impairments.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly patients without significant moderate to severe systemic comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Pulse Pressure Variation | Before induction
  PPV in tidal and during forced inspiratory breathing

SECONDARY OUTCOMES:
Systolic Pressure Variation | Before induction
  SPV in tidal and during forced inspiratory breathing
blood pressure | before and after induction
  SBP、DBP and MAP

CONTACTS AND LOCATIONS:
Overall Officials: Zhang wenjie, master, Principal Investigator — Department of Pain Management, Second Xiangya Hospital, Central South University, Changsha